CLINICAL TRIAL: NCT00106808
Title: A Phase 3, Randomized, Double-blind, Active Controlled, Multicenter Trial to Evaluate the Safety and Efficacy of Muraglitazar (BMS-298585) Compared to Pioglitazone in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control
Brief Title: Study of Muraglitazar Versus Pioglitazone in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV168-062
Record Dates: First submitted 2005-03-31; First posted 2005-04-01 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2007-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — muraglitazar; Pioglitazone

INTERVENTIONS:
Drug: Muraglitazar
Drug: Pioglitazone

SUMMARY:
The purpose of this study is to compare Muraglitazar and Pioglitazone in patients with Type 2 Diabetes. Both the safety and blood sugar lowering effects of these treatments will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* HbA1c > = 8.0% and < = 12.0%
* Serum triglyceride concentration < = 600 mg/dL
* Fasting c-peptide > = 1.0 ng/ml
* Body mass index < = 41 kg/m2
* Drug naive patients

Exclusion Criteria:

* History of MI (myocardial infarction), coronary angioplasty or bypass graft(s), valvular disease or repair, unstable angina pectoris, transient ischemic attack (TIA), cerebrovascular accidents, accelerated/malignant hypertension, or hypertension related CHF (congestive heart failure) within six months prior to screening and during the Lead-In Phase.
* Women of child Bearing Potential
* Uncontrolled hypertension, CHF defined as New York Heart Association (NYHA) Class II, III and IV, exacerbation of previously stable CHF (any NYHA class) or uncontrolled cardiac arrhythmia in the 30 days prior to screening and during the Lead-In Phase.
* History of renal disease, bladder cancer, pulmonary disease, gastrointestinal disease, active liver disease or endocrine disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440
Dates: Start 2005-08; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Change in HBA1c from baseline to Week 24

SECONDARY OUTCOMES:
Change for baseline in TG and HDL-C at Week 24
Change from baseline in FPG, fasting insulin, fasting c-peptide, body mass index, body weight, waist circumferance, SBP and DBP.
To assess safety and tolerability of both Muraglitazar regimens relative to pioglitazone regimen when administered for up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (195):
- United States (112):
  - Local Institution, Birmingham, Alabama
  - Local Institution, Columbiana, Alabama
  - Local Institution, Madison, Alabama
  - Local Institution, Glendale, Arizona
  - Local Institution, Mesa, Arizona
  - Local Institution, Peoria, Arizona
  - Local Institution, Phoenix, Arizona
  - Local Institution, Scottsdale, Arizona
  - Local Institution, Beverly Hills, California
  - Local Institution, Concord, California
  - Local Institution, Encinitas, California
  - Local Institution, Fresno, California
  - Local Institution, La Jolla, California
  - Local Institution, Los Angeles, California
  - Local Institution, Los Gatos, California
  - Local Institution, Orange, California
  - Local Institution, Pasadena, California
  - Local Institution, Roseville, California
  - Local Institution, Santa Monica, California
  - Local Institution, Colorado Springs, Colorado
  - Local Institution, Wilmington, Delaware
  - Local Institution, Boynton Beach, Florida
  - Local Institution, Charlotte Harbour, Florida
  - Local Institution, Chipley, Florida
  - Local Institution, Destin, Florida
  - Local Institution, Holly Hill, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Miami, Florida
  - Local Institution, New Port Richey, Florida
  - Local Institution, Niceville, Florida
  - Local Institution, Panama City, Florida
  - Local Institution, Port Charlotte, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Blue Ridge, Georgia
  - Local Institution, Calhoun, Georgia
  - Local Institution, Carrollton, Georgia
  - Local Institution, Dunwoody, Georgia
  - Local Institution, Marietta, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, North Chicago, Illinois
  - Local Institution, Evansville, Indiana
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Shawnee Mission, Kansas
  - Local Institution, Wichita, Kansas
  - Local Institution, Louisville, Kentucky
  - Local Institution, Lafayette, Louisiana
  - Local Institution, Shreveport, Louisiana
  - Local Institution, Baltimore, Maryland
  - Local Institution, Cantonville, Maryland
  - Local Institution, Towson, Maryland
  - Local Institution, Westminister, Maryland
  - Local Institution, Swansea, Massachusetts
  - Local Institution, Cadillac, Michigan
  - Local Institution, Portage, Michigan
  - Local Institution, Richland, Michigan
  - Local Institution, Gulfport, Mississippi
  - Local Institution, Tupelo, Mississippi
  - Local Institution, City of Saint Peters, Missouri
  - Local Institution, Excelsior Springs, Missouri
  - Local Institution, Butte, Montana
  - Local Institution, Missoula, Montana
  - Local Institution, Bridgewater, New Jersey
  - Local Institution, Cherry Hill, New Jersey
  - Local Institution, Binghamton, New York
  - Local Institution, Johnson City, New York
  - Local Institution, Mineola, New York
  - Local Institution, Northport, New York
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Greenville, North Carolina
  - Local Institution, Hickory, North Carolina
  - Local Institution, Morehead City, North Carolina
  - Local Institution, Salisbury, North Carolina
  - Local Institution, Wilmington, North Carolina
  - Local Institution, Barberton, Ohio
  - Local Institution, Bellbrook, Ohio
  - Local Institution, Canal Fulton, Ohio
  - Local Institution, Canfield, Ohio
  - Local Institution, Canton, Ohio
  - Local Institution, Columbus, Ohio
  - Local Institution, Lyndhurst, Ohio
  - Local Institution, Mentor, Ohio
  - Local Institution, Youngstown, Ohio
  - Local Institution, Eugene, Oregon
  - Local Institution, Medford, Oregon
  - Local Institution, Portland, Oregon
  - Local Institution, Philipsburg, Pennsylvania
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Reading, Pennsylvania
  - Local Institution, Tipton, Pennsylvania
  - Local Institution, West Grove, Pennsylvania
  - Local Institution, East Providence, Rhode Island
  - Local Institution, Greer, South Carolina
  - Local Institution, Mt. Pleasant, South Carolina
  - Local Institution, Simpsonville, South Carolina
  - Local Institution, Chattanooga, Tennessee
  - Local Institution, Fayetteville, Tennessee
  - Local Institution, Memphis, Tennessee
  - Local Institution, Selmer, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Corpus Christi, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Irving, Texas
  - Local Institution, Midland, Texas
  - Local Institution, New Braunfels, Texas
  - Local Institution, Pearland, Texas
  - Local Institution, Rosenberg, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Bountiful, Utah
  - Local Institution, Falls Church, Virginia
  - Local Institution, Norfolk, Virginia
  - Local Institution, Salem, Virginia
  - Local Institution, Spokane, Washington
- Argentina (5):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Chacabuco, Chaco Province
  - Local Institution, Corrientes, Corrientes Province
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Santa Fe, Santa Fe Province
- Australia (12):
  - Local Institution, Broadmeadow, New South Wales
  - Local Institution, Concord, New South Wales
  - Local Institution, Randwick, New South Wales
  - Local Institution, Westmead, New South Wales
  - Local Institution, Brisbane, Queensland
  - Local Institution, Cairns, Queensland
  - Local Institution, Daw Park, South Australia
  - Local Institution, Box Hill, Victoria
  - Local Institution, Fitzroy, Victoria
  - Local Institution, Geelong, Victoria
  - Local Institution, Melbourne, Victoria
  - Local Institution, Freemantle, Western Australia
- Brazil (8):
  - Local Institution, B. Rodolfo Teofilo, Ceará
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Cerq. Cesar, São Paulo
  - Local Institution, Guama, São Paulo
  - Local Institution, Paulistânia, São Paulo
  - Local Institution, Rua Maestro, São Paulo
  - Local Institution, Ruo Maestro Cardim, São Paulo
  - Local Institution, Vila Mariana, São Paulo
- Canada (18):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Coquitlam, British Columbia
  - Local Institution, Langley, British Columbia
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Antigonish, Nova Scotia
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Cambridge, Ontario
  - Local Institution, Kitchener, Ontario
  - Local Institution, London, Ontario
  - Local Institution, Markham, Ontario
  - Local Institution, North Bay, Ontario
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Windsor, Ontario
  - Local Institution, Greenfield Park, Quebec
  - Local Institution, Laval, Quebec
  - Local Institution, Longueuil, Quebec
- Local Institution, Santiago, Región de Valparaíso, Chile
- India (7):
  - Local Institution, Bangalore
  - Local Institution, Chennai
  - Local Institution, Hyderabad
  - Local Institution, Kolkata
  - Local Institution, Mumbai
  - Local Institution, New Delhi
  - Local Institution, Vellore
- Mexico (7):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Chihuahua City, Chihuahua
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Morelia, Michioacan
  - Local Institution, Monterrey, Nuevo León
- Local Institution, Lima, Peru
- Philippines (6):
  - Local Institution, Cebu
  - Local Institution, Las Piñas
  - Local Institution, Manila
  - Local Institution, Pasig
  - Local Institution, Quezon
  - Local Institution, Quezon City
- Russia (5):
  - Local Institution, Kirov
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
  - Local Institution, Yaroslavl
- Taiwan (3):
  - Local Institution, Kaohsiung City
  - Local Institution, Taipei
  - Local Institution, Taoyuan Hsien
- Thailand (4):
  - Local Institution, Bangkok
  - Local Institution, Kong Kaen
  - Local Institution, Songkhla
  - Local Institution, Taipei City
- Ukraine (6):
  - Local Institution, Dniepropetrovsk
  - Local Institution, Kharkiv
  - Local Institution, Kiev
  - Local Institution, Kyiv
  - Local Institution, Odesa
  - Local Institution, Simferopol